CLINICAL TRIAL: NCT05203796
Title: A Single-centered, Double-blinded, Placebo/Sham-controlled, Randomized Exploratory Clinical Trial to Evaluate the Transcutaneous Electrical Stimulation Medical Device's Safety and Effectiveness in Treating the Patients With Mild- or Moderate-level Dry Eye Disease Using NuEyne 02 (Personal Stimulator)
Brief Title: The Evaluation of the Transcutaneous Electrical Stimulation Medical Device's Safety and Effectiveness in Treating the Patients With Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE_DED_002
Record Dates: First submitted 2021-12-16; First posted 2022-01-24 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Dry eye disease patients (n=12) (Experimental): Patient needs to visit site at least 7 times(Screening, Baseline, wk1, wk2, wk3, wk4, wk5). From baseline visit, patients wear our clinical trial device 30mins per day for 5wks(2Hz stimulation). All other procedures during clinical trial the are the same.
  Intervention: Device: Transcutaneous pulsed electrical stimulation
  Interventions: Device: Transcutaneous pulsed electrical stimulation (NuEyne 02)
- Comparison group: Dry eye disease patients (n=12) (Sham Comparator): Patient needs to visit site at least 7 times(Screening, Baseline, wk1, wk2, wk3, wk4, wk5). From baseline visit, patients wear our clinical trial device 30mins per day for 5wks(sham stimulation). All other procedures during clinical trial the are the same.
  Intervention: Device: Sham device
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous pulsed electrical stimulation (NuEyne 02) — Arm 1: Experimental: Experimental group: Dry eye disease patients (n=12) Device: Pulse Electrical Stimulation Pulse Electrical Stimulation: Patients wear our clinical trial device 30mins once a day for 4 weeks.
  Arms: Experimental group: Dry eye disease patients (n=12)
Device: Sham stimulation — Arm 2: Sham Comparator: Comparison group: Dry eye disease patients (n=12) Device: Sham stimulation Sham stimulation: Patients wear our clinical trial device 30mins once a day for 4 weeks.
  Arms: Comparison group: Dry eye disease patients (n=12)

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness for applying the electrical stimulation transcutaneously around the eyes and peripheral nerves nearby. The outcomes are compared between the patients with mild- or moderate-level dry eye disease using the real electrical stimulator and the sham electrical stimulator.

DETAILED DESCRIPTION:
Duration of study period(per participant): Screening period (0-4weeks), Intervention period (5weeks).

Patient needs to visit site at least 3 times (Screening, V4, V6), V2 can be done with screening visit.

The clinical trial device performs a personal electrical stimulator around the eyes and peripheral nerves for 28 days (7 times/week, 30 minutes each time).

During the study period, dry eye examination and treatment methods (only eye drops provided in clinical trials are applied) are carried out in the same way.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 19 to 70 years old
* Those who are diagnosed with dry eyes at the time of screening and have complained of dry eyes, discomfort, foreign body sensation, pain, and changes in vision for more than three months.
* Patients with OSDI score of 23 or more
* Patients with Fluorescein corneal staining score of 4 or more
* Schirmer test I result is less than 10mm for 5 minutes
* TBUT (Tear film break up time) test result of less than 10 seconds
* Those who agree not to use eye drops other than artificial tears provided in this clinical trial during the clinical trial period
* A person who voluntarily agreed to participate in this clinical trial

Exclusion Criteria:

* Those who participated in other clinical trials within 30 days of screening.
* Those who applied medical devices to treat dry eye syndrome and IPL medication such as cyclosporin for treatment of dry eye syndrome and local steroid eye drops within one month from the screening date.
* Those who have worn contact lenses within 72 hours prior to screening or need to wear contact lenses during the clinical trial period
* Patients with a history of ophthalmic surgery within 3 months before screening.
* Those with a history of vision correction surgery (LASIK, LASEK), etc. within 6 months from the screening date
* Patients who received a lacrimal punctual occlusion or a tear point cauterization of the within 90 days of screening.
* Patients with symptoms of anterior uveitis or active blepharitis.
* Patients currently receiving treatment for allergic eye disease
* Patients with an abnormality of the eyelid structure
* Patients with moderate to severe meibomian gland disorders
* Those with underlying diseases such as glaucoma, burns, Steven Johnson Syndrome, vitamin A deficiency-related diseases, thyroid dysfunction-related diseases, and neurotropic keratinis.
* Other clinically significant ophthalmic diseases that are not caused by dry eye disease After corneal transplant surgery, corneal surface disease, abnormal corneal sensitivity, abnormal tear excess, etc. may confuse the interpretation of clinical trial results.
* Patients with uncontrolled systemic chronic diseases such as diabetes) or a history of malignant tumors
* Autoimmune disease patients
* People taking medications such as Steroids, immunosuppressants, omega 3 and anticholinergic drugs, etc.
* Pregnant or lactating women
* Among female subjects of childbearing potential, those who do not consent to contraception by a medically accepted method during this clinical trial period
* Medically permitted contraceptive methods: condoms, oral contraceptives that last at least three months, injections or insertion contraceptives, and installation of intrauterine contraceptives, etc.
* Patients with a history of drug or alcohol abuse
* People who are allergic to medicines such as Fluorescein Solution or eye drop anesthetics
* A person who is judged to have a problem in electrode attachment due to an inflammatory reaction or other dermatological problems in the periorbital skin where the electrode of the medical device for clinical trial is attached
* A person who is judged to have other reasons for prohibiting the use of medical devices for clinical trials
* Any other cases that PI considers hard to participate in this clinical trial(e.g. heart-related problems, seizure, epilepsy. Patients transplanted metal or electronic device in head & neck. Patient suffering from unknown pain. Patients who are warned not to use out clinical trial device or is prohibited from using it.)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Changes in Tear Break-Up Time(TBUT) | baseline, 2, 4 weeks
  Check the change of Tear Break-Up Time(TBUT) in the baseline, 2, 4 weeks
Changes in Corneal & Conjunctival Fluorescein staining score | baseline, 2, 4 weeks
  Check the change of Corneal & Conjunctival Fluorescein staining score in the baseline, 2, 4 weeks

SECONDARY OUTCOMES:
Changes in Ocular Surface Disease Index Dry Eye Questionnaires(OSDI) score | baseline, 2, 4 weeks
  Check the change of Ocular Surface Disease Index Dry Eye Questionnaires(OSDI) score in the baseline, 2, 4 weeks
Changes in A Five-item Dry Eye Questionnaire(DEQ-5) score | baseline, 2, 4 weeks
  Check the change of A Five-item Dry Eye Questionnaire(DEQ-5) score in the baseline, 2, 4 weeks
Changes in Visual Analog Scale(VAS) score | baseline, 2, 4 weeks
  Check the change of Visual Analog Scale(VAS) score in the baseline, 2, 4 weeks
Changes in Matrix Metalloproteinases-9(MMP-9) level | baseline, 2, 4 weeks
  Check the change of Matrix Metalloproteinases-9(MMP-9) level in the baseline, 2, 4 weeks
Changes in Tear Lipid Layer Thickness as measured by Lipiview | baseline, 2, 4 weeks
  Check the change of Tear Lipid Layer Thickness as measured by Lipiview in the baseline, 2, 4 weeks
Changes in Tear Volume as measured by Schirmer's Test | baseline, 2, 4 weeks
  Check the change of Tear Volume as measured by Schirmer's Test in the baseline, 2, 4 weeks
Changes in Tear Osmolarity | baseline, 2, 4 weeks
  Check the change of Tear Osmolarity in the baseline, 2, 4 weeks
Changes in Corneal Sensitivity as measured by aesthesiometer | baseline, 2, 4 weeks
  Check the change of Corneal Sensitivity as measured by aesthesiometer in the baseline, 2, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donghui Lim, Ph. D., MD., Principal Investigator — donghui.lim@samsung.com
Locations (1):
- Department of Ophthalmology, Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No